CLINICAL TRIAL: NCT07405307
Title: Evaluation of the Proportion of Patients With Gastrointestinal Cancer Who Have Symptoms of Sarcopenia
Brief Title: Sarcopenia Risk Screening in Patients With Gastrointestinal Cancer Using SARC-F
Status: Recruiting | Type: Observational
Sponsor: Institute of Oncology Ljubljana (Other)
Responsible Party: Sponsor
Other Study IDs: OIL-SARC-2023
Record Dates: First submitted 2026-02-04; First posted 2026-02-12 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Gastrointestinal Cancer; Sarcopenia
Keywords: SARC-F; sarcopenia screening; muscle mass loss
MeSH Terms: conditions — Gastrointestinal Neoplasms; Sarcopenia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Gastrointestinal Cancer Patients: Patients with gastrointestinal cancer receiving systemic treatment (adjuvant or metastatic setting) at the Institute of Oncology Ljubljana. Participants will be screened for sarcopenia risk using the SARC-F questionnaire at baseline and during treatment.
  Interventions: Other: Sarcopenia Screening and Nutritional Referral

INTERVENTIONS:
Other: Sarcopenia Screening and Nutritional Referral — Participants with a positive SARC-F screening result will be referred to the Clinical Nutrition Outpatient Clinic for further assessment of sarcopenia using anthropometric measurements and DXA, and for implementation of multidisciplinary interventions according to standard clinical practice.

SUMMARY:
Sarcopenia is a syndrome characterized by progressive loss of skeletal muscle mass and strength and is associated with worse outcomes in cancer patients. It can negatively affect prognosis, increase postoperative complications, reduce tolerance to systemic therapy, and impair quality of life. Sarcopenia may be present even in patients with preserved nutritional status or overweight.

This study aims to evaluate the proportion of patients with gastrointestinal cancer who are at risk of sarcopenia, as assessed by the SARC-F screening questionnaire, before initiation of systemic treatment and during treatment. Patients with a positive screening result may be referred for further nutritional evaluation and assessment of sarcopenia severity using anthropometric measurements and DXA, according to standard clinical practice.

DETAILED DESCRIPTION:
Sarcopenia is a complex condition characterized by progressive and generalized loss of skeletal muscle mass and strength. In oncology patients, sarcopenia is associated with increased mortality, higher rates of postoperative complications, reduced response to systemic therapy, increased treatment-related toxicity, and decreased quality of life. Sarcopenia may occur independently of malnutrition and may also be present in patients with normal or increased body weight.

Sarcopenia is not only related to the presence of malignant disease but may also develop or worsen as a consequence of oncological treatment. Several antineoplastic therapies have been shown to negatively affect muscle mass and function.

Due to its significant negative clinical impact, early detection of sarcopenia risk is essential. The SARC-F questionnaire is a validated screening tool recommended by the European Working Group on Sarcopenia in Older People (EWGSOP2) for identifying individuals at risk of sarcopenia.

This interventional study will evaluate the proportion of patients with gastrointestinal cancers treated at the Institute of Oncology Ljubljana who screen positive for sarcopenia risk using the SARC-F questionnaire before initiation of systemic treatment and during treatment. The study will also assess changes in the proportion of patients at risk over time.

Patients with a positive SARC-F screening result may be referred to the clinical nutrition outpatient clinic for further evaluation, including anthropometric measurements and DXA assessment, in order to determine the severity of sarcopenia. Based on clinical evaluation and in agreement with the treating oncologist, multimodal and multidisciplinary preventive and therapeutic interventions may be introduced as part of routine clinical care.

The study duration is planned for two years.

ELIGIBILITY:
Inclusion Criteria:

Adult patients (≥18 years) with gastrointestinal cancer

Patients planned for or receiving systemic anticancer treatment (adjuvant treatment or treatment of metastatic disease)

Ability to complete the SARC-F screening questionnaire

Written informed consent provided

Exclusion Criteria:

Patients younger than 18 years

Patients unable to complete the questionnaire (e.g., severe cognitive impairment or inability to cooperate)

Patients not eligible for systemic anticancer treatment

Refusal to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with gastrointestinal cancers treated at the Institute of Oncology Ljubljana, receiving systemic therapy either in the adjuvant setting or for metastatic disease. Patients will be screened for sarcopenia risk using the SARC-F questionnaire before treatment initiation and during systemic therapy.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of gastrointestinal cancer patients with positive SARC-F screening | Baseline (before start of systemic treatment) and during systemic treatment (after 3 months
  Percentage of patients with gastrointestinal cancer who screen positive for sarcopenia risk using the SARC-F questionnaire. A SARC-F score ≥4 will be considered positive.

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Oncology Ljubljana, Ljubljana, Slovenia

IPD SHARING:
Plan to Share IPD: No